CLINICAL TRIAL: NCT02074319
Title: A Randomised Double Blind Placebo Controlled 12 Week Trial of Methotrexate Added to Treatment As Usual in Early Schizophrenia
Brief Title: RCT of Methotrexate Added to Treatment As Usual in Schizophrenia
Acronym: RECOVERY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Abbasi Shaheed Hospital (Other); Dow University of Health Sciences (Other); Karwan e Hayat, Karachi, Pakistan (Unknown); Institute of Behavioural Sciences, Karachi, Pakistan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RECOVERY-001
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Anti-Inflammatory; Methotrexate; Psychosis Not Otherwise Specified
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo for methotrexate
  Interventions: Drug: Methotrexate
- Methotrexate (Experimental): Methotrexate 10 mg once a week orally
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Treatment as usual or standard treatment for psychosis will be common in all arms

SUMMARY:
The aim of the this study is to evaluate the effectiveness of methotrexate added to treatment as usual on positive and negative symptoms, cognitive and social functioning and quality of life of patients suffering from schizophrenia.

DETAILED DESCRIPTION:
The purpose of the study is to test the prediction that addition of methotrexate to treatment as usual (TAU) for patients with schizophrenia will result in following outcomes:

* Primary:

  * improvement in negative symptoms
  * improvement in positive symptoms
* Secondary:

  * improvement in social functioning
  * improvement in cognitive functions
  * acceptability and tolerability of methotrexate added to TAU A total 72 participants (36 participants in intervention group and 36 in control group) meeting inclusion criteria of the study will be recruited and randomized in study in two arms. Research assistants and participating psychiatrists will assess participants for eligibility criteria. After providing detailed information regarding study by using patient information sheet, written informed consent will be taken from participants. Trained research assistant will asses participants at baseline, 2, 4, 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, indicating that the subject understood the purpose of and procedures required for the study, before the initiation of any study specific procedures
* Aged 18 to 35 years
* Diagnostic and Statistical Manual-IV (DSM-IV) diagnosed first episode psychosis, schizophrenia, schizoaffective disorder, psychosis not otherwise specified or schizophreniform disorder.
* First episode (within first 5 years of diagnosis)
* Competent and willing to give informed consent
* Medication remained stable 4 weeks prior to baseline.
* Able to take oral medication and likely to complete the required evaluations.
* Female participants of child bearing capability must be willing to use adequate contraceptives for the duration of the study, and, willing to have a pregnancy test pre treatment and at ten weekly intervals while on study medication.

  1. Adequate contraception is defined as use of contraceptive double barrier system (i.e. condom and spermicide) or contraceptive implant, oral contraceptive or injected depot contraceptive plus other form of contraceptive i.e. condom. Females will be considered incapable of child bearing if they are one year post-menopausal or irreversibly surgically sterilised.

Exclusion Criteria:

* Violation of any inclusion criteria
* Failure to perform screening or baseline examinations
* Relevant ICD 10 organic brain disease or neurological diagnoses
* Patients with liver disease
* Patients who will meet the criteria for a DSM-IV TR diagnosis of alcohol or substance abuse (other than for nicotine) within the last month or the criteria for DSM-IV TR alcohol or substance dependence (other than for nicotine) within the last 6 months
* Any change of psychotropic medications within the previous 4 weeks
* Recreational drugs or alcohol abuse
* Pregnant or lactating women and those of reproductive age without adequate contraception
* Relevant medical illness will be determined in the first instance by asking the patients mental health care team if the patient has any medical condition/problems. After consent has been obtained the research nurse/ research doctor will then have access to the patients' notes and will assess patient eligibility to take part in the clinical trial by scrutinising the patients' past medical history, most recent blood results, electrocardiograms, as well as any physical tests that have been performed on the patient.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale PANSS | 3 months
  PANSS is an assessment measures to assess severity of symptoms of schizophrenia

SECONDARY OUTCOMES:
CogState | 3 months
  Measuring all seven domains recommended by MATRICS (NIMH initiative). These domains include speed processing, attention/vigilance, Working memory (nonverbal & verbal), verbal learning, visual learning, reasoning and problem solving and social cognitions.

OTHER OUTCOMES:
Social Functioning Scale | 3 months
  Self-rating questionnaire assessing social functioning in 7 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Imran B Chaudhry, MD, Principal Investigator — University of Manchester
Locations (4):
- Pakistan (4):
  - Abasi Shaheed Hospital, Karachi, Sindh
  - Civil hospital Karachi, Karachi, Sindh
  - Institute of Behavioural Sciences, Karachi, Sindh
  - Karwn e Hayat, Karachi, Sindh

REFERENCES:
- [Background] Chaudhry IB, Hallak J, Husain N, Minhas F, Stirling J, Richardson P, Dursun S, Dunn G, Deakin B. Minocycline benefits negative symptoms in early schizophrenia: a randomised double-blind placebo-controlled clinical trial in patients on standard treatment. J Psychopharmacol. 2012 Sep;26(9):1185-93. doi: 10.1177/0269881112444941. Epub 2012 Apr 23. PMID 22526685
- [Background] Behrens MM, Ali SS, Dugan LL. Interleukin-6 mediates the increase in NADPH-oxidase in the ketamine model of schizophrenia. J Neurosci. 2008 Dec 17;28(51):13957-66. doi: 10.1523/JNEUROSCI.4457-08.2008. PMID 19091984
- [Background] Bernstein HG, Steiner J, Bogerts B. Glial cells in schizophrenia: pathophysiological significance and possible consequences for therapy. Expert Rev Neurother. 2009 Jul;9(7):1059-71. doi: 10.1586/ern.09.59. PMID 19589054
- [Background] Busse S, Busse M, Schiltz K, Bielau H, Gos T, Brisch R, Mawrin C, Schmitt A, Jordan W, Muller UJ, Bernstein HG, Bogerts B, Steiner J. Different distribution patterns of lymphocytes and microglia in the hippocampus of patients with residual versus paranoid schizophrenia: further evidence for disease course-related immune alterations? Brain Behav Immun. 2012 Nov;26(8):1273-9. doi: 10.1016/j.bbi.2012.08.005. Epub 2012 Aug 14. PMID 22917959
- [Background] Cronstein BN. Low-dose methotrexate: a mainstay in the treatment of rheumatoid arthritis. Pharmacol Rev. 2005 Jun;57(2):163-72. doi: 10.1124/pr.57.2.3. PMID 15914465
- [Background] Doorduin J, de Vries EF, Willemsen AT, de Groot JC, Dierckx RA, Klein HC. Neuroinflammation in schizophrenia-related psychosis: a PET study. J Nucl Med. 2009 Nov;50(11):1801-7. doi: 10.2967/jnumed.109.066647. Epub 2009 Oct 16. PMID 19837763
- [Background] Drzyzga L, Obuchowicz E, Marcinowska A, Herman ZS. Cytokines in schizophrenia and the effects of antipsychotic drugs. Brain Behav Immun. 2006 Nov;20(6):532-45. doi: 10.1016/j.bbi.2006.02.002. Epub 2006 Apr 3. PMID 16580814
- [Background] Godfrey PS, Toone BK, Carney MW, Flynn TG, Bottiglieri T, Laundy M, Chanarin I, Reynolds EH. Enhancement of recovery from psychiatric illness by methylfolate. Lancet. 1990 Aug 18;336(8712):392-5. doi: 10.1016/0140-6736(90)91942-4. PMID 1974941
- [Background] Gong K, Zhang Z, Sun X, Zhang X, Li A, Yan J, Luo Q, Gao Y, Feng Y. The nonspecific anti-inflammatory therapy with methotrexate for patients with chronic heart failure. Am Heart J. 2006 Jan;151(1):62-8. doi: 10.1016/j.ahj.2005.02.040. PMID 16368293
- [Background] Johnston A, Gudjonsson JE, Sigmundsdottir H, Ludviksson BR, Valdimarsson H. The anti-inflammatory action of methotrexate is not mediated by lymphocyte apoptosis, but by the suppression of activation and adhesion molecules. Clin Immunol. 2005 Feb;114(2):154-63. doi: 10.1016/j.clim.2004.09.001. PMID 15639649
- [Background] Mansur RB, Zugman A, Asevedo EM, da Cunha GR, Bressan RA, Brietzke E. Cytokines in schizophrenia: possible role of anti-inflammatory medications in clinical and preclinical stages. Psychiatry Clin Neurosci. 2012 Jun;66(4):247-60. doi: 10.1111/j.1440-1819.2012.02354.x. PMID 22624729
- [Background] Miller BJ, Buckley P, Seabolt W, Mellor A, Kirkpatrick B. Meta-analysis of cytokine alterations in schizophrenia: clinical status and antipsychotic effects. Biol Psychiatry. 2011 Oct 1;70(7):663-71. doi: 10.1016/j.biopsych.2011.04.013. Epub 2011 Jun 8. PMID 21641581
- [Background] Monji A, Kato T, Kanba S. Cytokines and schizophrenia: Microglia hypothesis of schizophrenia. Psychiatry Clin Neurosci. 2009 Jun;63(3):257-65. doi: 10.1111/j.1440-1819.2009.01945.x. PMID 19579286
- [Background] Morgan SL, Baggott JE, Vaughn WH, Austin JS, Veitch TA, Lee JY, Koopman WJ, Krumdieck CL, Alarcon GS. Supplementation with folic acid during methotrexate therapy for rheumatoid arthritis. A double-blind, placebo-controlled trial. Ann Intern Med. 1994 Dec 1;121(11):833-41. doi: 10.7326/0003-4819-121-11-199412010-00002. PMID 7978695
- [Background] Myint AM. Kynurenines: from the perspective of major psychiatric disorders. FEBS J. 2012 Apr;279(8):1375-85. doi: 10.1111/j.1742-4658.2012.08551.x. Epub 2012 Mar 27. PMID 22404766
- [Background] Potvin S, Stip E, Sepehry AA, Gendron A, Bah R, Kouassi E. Inflammatory cytokine alterations in schizophrenia: a systematic quantitative review. Biol Psychiatry. 2008 Apr 15;63(8):801-8. doi: 10.1016/j.biopsych.2007.09.024. Epub 2007 Nov 19. PMID 18005941
- [Background] Procter A. Enhancement of recovery from psychiatric illness by methylfolate. Br J Psychiatry. 1991 Aug;159:271-2. doi: 10.1192/bjp.159.2.271. PMID 1773245
- [Background] Rajagopalan PT, Zhang Z, McCourt L, Dwyer M, Benkovic SJ, Hammes GG. Interaction of dihydrofolate reductase with methotrexate: ensemble and single-molecule kinetics. Proc Natl Acad Sci U S A. 2002 Oct 15;99(21):13481-6. doi: 10.1073/pnas.172501499. Epub 2002 Oct 1. PMID 12359872
- [Background] Schulte-Herbruggen O, Nassenstein C, Lommatzsch M, Quarcoo D, Renz H, Braun A. Tumor necrosis factor-alpha and interleukin-6 regulate secretion of brain-derived neurotrophic factor in human monocytes. J Neuroimmunol. 2005 Mar;160(1-2):204-9. doi: 10.1016/j.jneuroim.2004.10.026. Epub 2004 Dec 22. PMID 15710474
- [Background] van Berckel BN, Bossong MG, Boellaard R, Kloet R, Schuitemaker A, Caspers E, Luurtsema G, Windhorst AD, Cahn W, Lammertsma AA, Kahn RS. Microglia activation in recent-onset schizophrenia: a quantitative (R)-[11C]PK11195 positron emission tomography study. Biol Psychiatry. 2008 Nov 1;64(9):820-2. doi: 10.1016/j.biopsych.2008.04.025. Epub 2008 Jun 4. PMID 18534557
- [Background] Whittle SL, Hughes RA. Folate supplementation and methotrexate treatment in rheumatoid arthritis: a review. Rheumatology (Oxford). 2004 Mar;43(3):267-71. doi: 10.1093/rheumatology/keh088. Epub 2004 Jan 6. PMID 14963199
- [Background] Zhang Z, Zhao P, Li A, Lv X, Gao Y, Sun H, Ding Y, Liu J. Effects of methotrexate on plasma cytokines and cardiac remodeling and function in postmyocarditis rats. Mediators Inflamm. 2009;2009:389720. doi: 10.1155/2009/389720. Epub 2009 Oct 26. PMID 19884981
- [Derived] Chaudhry IB, Husain N, ur Rahman R, Husain MO, Hamirani MM, Kazmi A, Baig S, Haddad PM, Buch MH, Qureshi I, Mehmood N, Kiran T, Fu B, Afsar S, Deakin B. A randomised double-blind placebo-controlled 12- week feasibility trial of methotrexate added to treatment as usual in early schizophrenia: study protocol for a randomised controlled trial. Trials. 2015 Jan 7;16:9. doi: 10.1186/1745-6215-16-9. PMID 25563714
- See also: Website of Pakistan Institute of Learning and Living — http://pill.org.pk